CLINICAL TRIAL: NCT00435825
Title: A Randomized, Double-blind Study of the Effect of Treatment Duration and Dose of PEGASYS on HBeAg Seroconversion and Safety in Patients With HBeAg Positive Chronic Hepatitis B.
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With Hepatitis Be Antigen (HBeAg) Positive Chronic Hepatitis B (CHB).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WV19432
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- peginterferon alfa-2a 90 μg_24 Weeks (Experimental): Participants received 90 micrograms (μg) peginterferon alfa-2a subcutaneous once a week for 24 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- peginterferon alfa-2a 180 μg_24 Weeks (Experimental): Participants received 180 μg peginterferon alfa-2a subcutaneous once a week for 24 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- peginterferon alfa-2a 90 μg_48 Weeks (Experimental): Participants received 90 μg peginterferon alfa-2a subcutaneous once a week for 48 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- peginterferon alfa-2a 180 μg_48 Weeks (Experimental): Participants received 180 μg peginterferon alfa-2a subcutaneous once a week for 48 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 90 or 180 micrograms subcutaneous weekly for 24 weeks or 48 weeks.

SUMMARY:
This 4 arm study will compare the efficacy and safety of PEGASYS given for 24 or 48 weeks, and at doses of 90 or 180 micrograms weekly, in the treatment of HBeAg positive patients with chronic hepatitis B. Patients will be randomized to one of 4 treatment groups: a)PEGASYS 90 micrograms subcutaneous (sc) weekly for 24 weeks, b)PEGASYS 180 micrograms sc weekly for 24 weeks, c)PEGASYS 90 micrograms sc weekly for 48 weeks or d)PEGASYS 180 micrograms sc weekly for 48 weeks. Following treatment there will be a 24 week period of treatment-free follow-up in all treatment groups for the primary endpoint. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* positive Hepatitis B surface antigen (HBsAg) for >6 months, positive HBeAg, HBV DNA >500,000 copies/mL, and anti-HBs negative;
* liver disease consistent with Chronic Hepatitis B.

Exclusion Criteria:

* antiviral therapy for CHB within previous 6 months;
* co-infection with Hepatitis A virus (HAV), Hepatitis C virus (HCV), Hepatitis D virus (HDV) or Human immuno deficiency virus (HIV);
* evidence of decompensated liver disease;
* medical condition associated with chronic liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- United States (10):
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Atlanta, Georgia
  - Flushing, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Richmond, Virginia
- Australia (3):
  - Fitzroy
  - Greenslopes
  - Woolloongabba
- Brazil (5):
  - Campinas
  - Ribeirão Preto
  - Salvador
  - Santo André
  - São Paulo
- China (4):
  - Beijing
  - Guangzhou
  - Hunan
  - Shanghai
- France (6):
  - Clichy
  - Montpellier
  - Nice
  - Strasbourg
  - Toulouse
  - Villejuif
- Germany (5):
  - Berlin
  - Cologne
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Hanover
- Hong Kong, Hong Kong
- New Zealand (2):
  - Auckland
  - Hamilton
- Russia (4):
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Songkhla

REFERENCES:
- [Derived] Liaw YF, Jia JD, Chan HL, Han KH, Tanwandee T, Chuang WL, Tan DM, Chen XY, Gane E, Piratvisuth T, Chen L, Xie Q, Sung JJ, Wat C, Bernaards C, Cui Y, Marcellin P. Shorter durations and lower doses of peginterferon alfa-2a are associated with inferior hepatitis B e antigen seroconversion rates in hepatitis B virus genotypes B or C. Hepatology. 2011 Nov;54(5):1591-9. doi: 10.1002/hep.24555. PMID 22045673

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Started | 141 | 136 | 138 | 136
Received Study Drug | 140 | 136 | 136 | 136
Entered Follow-up | 140 | 132 | 135 | 133
Completed 24 Weeks Treatment | 128 | 126 | 134 | 131
Completed 48 Weeks Treatment | 0 | 0 | 124 | 117
Completed | 123 (Completed is the number of participants who received study treatment and completed follow-up.) | 124 | 127 | 120
Not Completed | 18 | 12 | 11 | 16
Not completed — Abnormality of Laboratory Test | 0 | 1 | 0 | 0
Not completed — Insufficient Therapeutic Response | 3 | 1 | 0 | 3
Not completed — Other Protocol Violation | 1 | 0 | 0 | 0
Not completed — Refused treatment | 2 | 0 | 0 | 5
Not completed — Failure to return | 5 | 0 | 4 | 0
Not completed — Did not receive study drug | 1 | 0 | 2 | 0
Not completed — Did not enter follow-up | 0 | 4 | 1 | 3
Not completed — Did not complete full follow-up period | 6 | 6 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Measures are based on participants from the Intent-to-treat population who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks | Total
Number analyzed (Participants) | 140 | 136 | 136 | 136 | 548
Age, Customized [Mean (Full Range); unit: Years] | 31.8 (9.77) [18 to 56] | 33.0 (10.52) [18 to 66] | 33.8 (10.48) [16 to 62] | 33.3 (10.89) [18 to 69] | 32.98 [16 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 39 | 40 | 48 | 171
  Male | 96 | 97 | 96 | 88 | 377

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis Be Antigen (HBeAg) Seroconversion 24 Weeks Following End of Treatment
Description: Blood was collected for HBeAg. HBeAg seroconversion was defined as the absence of HBeAg (a negative result for HBeAg) and the presence of anti-HBe (a positive result for anti-HBe) determined at 24 weeks after the end of treatment.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: Per-protocol population defined as all participants who received study drug and who did not have any major protocol deviation. Patients were analyzed according to the treatment received, rather than the randomized treatment. 10 patients in the per-protocol population switched treatment groups for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 14.08 [8.82 to 20.91] | 22.86 [16.19 to 30.71] | 25.76 [18.54 to 34.09] | 36.15 [27.91 to 45.04]

2. Secondary Outcome: Percentage of Participants With Hepatitis Be Antigen (HBeAg) Seroconversion at Week 72
Description: Blood was collected for HBeAg. HBeAg seroconversion was defined as the absence of HBeAg (a negative result for HBeAg) and the presence of anti-HBe (a positive result for anti-HBs) determined at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 18.31 [12.32 to 25.67] | 27.14 [19.98 to 35.30] | 25.76 [18.54 to 34.09] | 36.15 [27.91 to 45.04]

3. Secondary Outcome: Percentage of Participants With Loss of Hepatitis Be Antigen (HBeAg) 24 Weeks Following End of Treatment
Description: Blood was collected HBeAg 24 Weeks following the end of treatment. Loss of HBeAg is defined as the absence of HBeAg.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: Per-protocol population defined as all participants who received study drug and who did not have any major protocol deviation. Patients were analyzed according to the treatment received, rather than the randomized treatment. 10 patients in the Per protocol population switched treatment groups for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 14.79 [9.39 to 21.71] | 22.86 [16.19 to 30.71] | 26.52 [19.21 to 34.90] | 36.15 [27.91 to 45.04]

4. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroconversion 24 Weeks Following the End of Treatment
Description: HBsAg seroconversion was defined as the absence of HBsAg (a negative result for HBsAg) and the presence of anti-HBs (a positive result for anti-HBs) determined at 24 weeks after the end of treatment.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 0.0 [0.0 to 2.56] | 0.0 [0.0 to 2.60] | 1.52 [0.18 to 5.37] | 2.31 [0.48 to 6.60]

5. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Surface Antigen (HBsAg) 24 Weeks Following End of Treatment
Description: Blood was collected for HBsAg 24 weeks following the end of treatment. Loss of HBsAg is defined as the absence of HBsAg.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 0.70 [0.02 to 3.86] | 0.0 [0.00 to 2.60] | 2.27 [0.47 to 6.50] | 2.31 [0.48 to 6.60]

6. Secondary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT)
Description: Blood was collected 24 weeks following the end of treatment for ALT and was analyzed at a local laboratory. A normal ALT is a value within the normal range of the assay.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 30.28 [22.86 to 38.55] | 30.71 [23.20 to 39.06] | 43.18 [34.59 to 52.08] | 52.31 [43.37 to 61.14]

7. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) Suppression < 20,000 IU/mL 24 Weeks Following End of Treatment
Description: Blood was collected for HBV-DNA 24 weeks following the end of treatment and was analyzed at the central laboratory using the Roche approved polymerase chain reaction (PCR) methodology. Percentage of participants with a HBV-DNA suppression of < 20,000 IU/mL (Less than 100,000 copies/mL) is reported.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 21.83 [15.34 to 29.53] | 21.43 [14.95 to 29.16] | 32.58 [24.68 to 41.27] | 42.31 [33.70 to 51.28]

8. Secondary Outcome: Percentage of Participants With Hepatitis Deoxyribonucleic Acid (HBV-DNA) Suppression < 2,000 IU/mL 24 Weeks Following End of Treatment
Description: Blood was collected for HBV-DNA and was analyzed at the central laboratories using the Roche approved PCR methodology 24 weeks following the end of treatment. Percentage of participants with A HBV-DNA Suppression of < 2,000 IU/mL (Less than 10,000 copies/mL) is reported.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment of Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 11.27 [6.58 to 17.65] | 11.43 [6.68 to 17.90] | 22.73 [15.89 to 30.83] | 30.0 [22.28 to 38.66]

9. Secondary Outcome: Percentage of Participants With Combined Endpoint Response 24 Weeks Following End of Treatment
Description: Combined endpoint was defined as HBeAg seroconversion, a normal serum ALT and HBV-DNA suppression below 20,000 IU/mL.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 7.75 [3.93 to 13.44] | 15.0 [9.53 to 22.01] | 17.42 [11.38 to 24.99] | 31.54 [23.67 to 40.27]

10. Secondary Outcome: Percentage of Participants With Dual Endpoint Response 24 Weeks Following End of Treatment
Description: Dual endpoint was defined as the achievement of both HBeAg seroconversion and a HBV-DNA <2,000 IU/ml (Less than 10,000 copies/mL).
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 142 | 140 | 132 | 130
Percentage of participants | 7.75 [3.93 to 13.44] | 9.29 [5.04 to 15.36] | 13.64 [8.29 to 20.69] | 24.62 [17.49 to 32.94]

11. Secondary Outcome: Quantitative Serum Alanine Aminotransferase (ALT) 24 Weeks Following End of Treatment
Description: Blood was collected 24 weeks following the end of treatment for ALT and was analyzed at a local laboratory. A normal ALT is a value within the normal range of the assay: 0- 55 units/liter (U/L).
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: Participants from the Per-protocol population defined as all participants who received study drug and who did not have any major protocol deviation who had data available for analysis. Patients were analyzed according to the treatment received. 10 patients in the per-protocol population switched treatment groups for the analysis.
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 131 | 133 | 126 | 124
U/L | 1.90 [1.84 to 1.96] | 1.97 [1.90 to 2.05] | 1.90 [1.82 to 1.98] | 1.73 [1.67 to 1.79]

12. Secondary Outcome: Quantitative HBV-DNA 24 Weeks Following End of Treatment
Description: Blood was collected for HBV-DNA and was analyzed at the central laboratories using the Roche approved PCR methodology 24 weeks following the end of treatment.
Time Frame: 24 Weeks following end of treatment (Week 48 for 24 Week Treatment or Week 72 for 48 Week Treatment)
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: IU/mL Log10
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Number analyzed (Participants) | 128 | 129 | 125 | 124
IU/mL Log10 | 6.33 [5.93 to 6.72] | 6.38 [5.99 to 6.76] | 5.98 [5.51 to 6.45] | 5.29 [4.81 to 5.78]

ADVERSE EVENTS:
Description: Safety set included randomized patients who received study drug and had at least 1 post-baseline assessment. 1 patient in the PEG-IFN 180 μg 24 week arm had no post-baseline assessments. 10 patients actually received drug for less time and switched arms for analysis (4 PEG-IFN 90 μg 48 weeks to 24 weeks and 6 PEG-IFN 180 μg 48 weeks to 24 weeks.
Arm/Group | Peginterferon Alfa-2a 90 μg_24 Weeks | Peginterferon Alfa-2a 180 μg_24 Weeks | Peginterferon Alfa-2a 90 μg_48 Weeks | Peginterferon Alfa-2a 180 μg_48 Weeks
Serious Adverse Events (participants affected / at risk) | 4/144 | 4/141 | 6/132 | 5/130
Other Adverse Events (participants affected / at risk) | 94/144 | 109/141 | 92/132 | 105/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 90 μg_24 Weeks (N=144) | Peginterferon Alfa-2a 180 μg_24 Weeks (N=141) | Peginterferon Alfa-2a 90 μg_48 Weeks (N=132) | Peginterferon Alfa-2a 180 μg_48 Weeks (N=130)
Hepatitis B (Infections and infestations) | 1 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 90 μg_24 Weeks (N=144) | Peginterferon Alfa-2a 180 μg_24 Weeks (N=141) | Peginterferon Alfa-2a 90 μg_48 Weeks (N=132) | Peginterferon Alfa-2a 180 μg_48 Weeks (N=130)
Pyrexia (General disorders) | 40 | 50 | 43 | 46
Fatigue (General disorders) | 27 | 20 | 29 | 32
Malaise (General disorders) | 1 | 9 | 8 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 24 | 26 | 41
Rash (Skin and subcutaneous tissue disorders) | 7 | 7 | 5 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 4 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 35 | 19 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 6 | 8
Headache (Nervous system disorders) | 23 | 35 | 23 | 25
Dizziness (Nervous system disorders) | 5 | 8 | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 7 | 14
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 6 | 10
Nausea (Gastrointestinal disorders) | 3 | 5 | 3 | 8
Nasopharyngitis (Infections and infestations) | 8 | 7 | 11 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 4 | 9
Insomnia (Psychiatric disorders) | 8 | 11 | 11 | 16
Decreased appetite (Metabolism and nutrition disorders) | 6 | 10 | 10 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.